CLINICAL TRIAL: NCT05986071
Title: A Phase I/II Study Evaluating M1774, an ATR Inhibitor, in Combination With Fulvestrant in Hormone Receptor-positive and HER2-negative, Advanced Breast Cancers, Resistant to CDK4/6 Inhibitor Plus Aromatase Inhibitor-based Endocrine Treatment
Brief Title: I/II Phase Study Evaluating M1774 in Combination With Fulvestrant in HR+ and HER2- Advanced Breast Cancers
Acronym: MATRIX
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: National Cancer Institute, France (Other Government); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MATRIx-IPC 2022-029
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: M1774; fulvestrant; CDK4/6; breast cancer; homologous recombination deficiency
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: Phase I : we will examine the safety and determine the recommended phase II dose (RP2D) of the combination of M1774 with Fulvestrant in ER+/HER2- ABC with progressive disease under or after CDK4/6 inhibitor and aromatase inhibitor.
  Phase II: Administration of M1774 ar RP2D with fulvestrant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): administration of M1774 in combination with fulvestrant
  Interventions: Drug: M1774; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: M1774 — • Phase I part = administration of M1774 in combination with fulvestrant in ER+/HER2- ABC resistant to CDK4/6 inhibitor and aromatase inhibitor-based endocrine therapy in order to detemine the recommended phase II dose Phase II part = administration of M1774 at RP2D in combination with fulvestrant
Drug: Fulvestrant injection — Phase I part = administration of M1774 in combination with fulvestrant in ER+/HER2- ABC resistant to CDK4/6 inhibitor and aromatase inhibitor-based endocrine therapy in order to detemine the recommended phase II dose Phase II part = administration of M1774 at RP2D in combination with fulvestrant

SUMMARY:
CDK4/6 inhibitor in combination with endocrine treatment is the standard of care in advanced breast cancer (ABC) with expression of hormone receptors and without HER2 overexpression (ER+/HER2-). When patients experience disease progression under this strategy, options of second-line endocrine treatment in combination with other targeted therapies are limited and have failed to improve overall survival to date over endocrine treatment alone. A significant fraction of ER+/HER2- ABC display genetic alterations associated with homologous recombination deficiency (HRD) which may be associated with efficacy of therapeutic targeting DNA damage response (DDR) pathways. Moreover, other molecular alterations associated with replicative stress may be found in ER+/HER2- ABC patients which may also favor antitumor activity of DDR targeting therapeutics. M1774 is a novel orally administered inhibitor of ataxia telangiectasia and rad3-related (ATR), a protein kinase with key activity in DDR pathway. MATRIx is a phase I/II study aiming to determine the recommended phase II dose (RP2D, phase I) as well as efficacy and safety (phase II) of M1774 in combination with fulvestrant in ER+/HER2-ABC patients whose disease has become resistant to aromatase inhibitor plus CDK4/6 inhibitor, and whose tumor displays molecular alterations associated with HRD, oncogenic driver activation and/or replicative stress. Primary endpoints will include: maximum tolerated dose (MTD) of M1774 in combination with fulvestrant (phase I), the clinical benefit rate and toxicity of the combination at RP2D of M1774 in the molecularly selected population (phase II). Baseline, on-treatment and post-treatment blood and tumor tissue samples will be collected for pharmacokinetics and translational analyses including genomic characterization of tumor tissue and ctDNA as well as functional studies focusing on DDR pathways.

DETAILED DESCRIPTION:
Approximately 5% among all types of breast cancers are associated with germline breast cancer susceptibility gene BRCA 1 or 2 mutations (gBRCA). These mutations lead to homologous recombination deficiency (HRD) and inability for cancer cells to repair DNA double-strand break (DDSB), making gBRCA-ABC exquisitely sensitive to poly(adenosine diphosphate-ribose) polymerase (PARP) inhibitors (22). Indeed, PARP is a pivotal actor in the repair of DNA single-strand breaks (DSSB), and PARP inhibition will generate accumulating DSSB leading to DDSB and ultimately cell death if let unrepaired, as it is in the context of HRD. In OlympiAD and EMBRACA trials assessing the efficacy of olaparib or talazoparib, respectively compared to physician's choice single-agent, non platin-based, chemotherapy in gBRCA HER2- ABC patients, a significant increase in PFS and an improvement in QOL was shown with both PARP inhibitors (23, 24) . Of note, around 50% of the patients in these trials had ER+/HER2- breast cancer. Among these patients the PFS was 7 month and 8.6 month with olaparib and talazoparib respectively. Yet, either in this subgroup or in the overall population, there was no OS improvement (25, 26). Nevertheless, according to guidelines (3), PARP inhibitors should be part of the treatment sequence in gBRCA, ER+ /HER2- ABC patients when the disease becomes resistant to CDK4/6 inhibitor-based first-line ET.

Even in the absence of gBRCA, HRD may still exist in tumors due to somatic defects in BRCA genes as well as alterations in other genes involved in homologous recombination repair such as ATM, BARD1, CHEK1, CHEK2, RAD51C, RAD51D, BRIP1, NBN, PALB2, and the Fanconi anemia complementation group (FANC) family of genes (FANCA, FANCC, FANCD2, FANCE, FANCF, FANCG, and FANCL): the so-called "BRCAness" phenotype (27). In whole-exome studies focusing on ABC samples, we and others found that more than approximately 15% of ER+/HER2- ABC may display such a BRCAness phenotype (28-30). Although it should be theoretically associated with similar sensitivity to PARP inhibitors, clinical data examining anti-tumor activity of this latter class remain relatively sparse. In a recent study investigating antitumor activity of olaparib in ABC with either germline mutations in HR-related genes other than BRCA1/2 or somatic BRCA1/2 mutations, only patients with gPALB2 or somatic BRCA mutations but not those with mutations in other homologous recombination-associated genes had high response rates and clinical benefit (31). Thus, developing alternative therapeutic targeting DNA damage response (DDR) pathways in BRCA and non BRCA-driven HRD is urgently needed.

DNA damage repair pathway :

The DDR pathway, which coordinates the detection of cellular DNA damage with cell-cycle adaptation and repair processes, primarily involves ataxia telangiectasia and rad3-related (ATR), ataxia telangiectasia mutated (ATM), and DNA-dependent protein kinase (DNA-PK/PRKDC). ATR, the key DDR kinase, is activated by accumulated DSSB, primarily induced by oncogene-driven dysregulated replication, leading to the so-called replication stress (RS) and associated genomic instability. Once activated, ATR phosphorylates checkpoint kinase 1 (CHK1), leading to cell-cycle arrest, pausing of DNA synthesis and initiation of DNA repair. Loss of ATR function leads to the inability to resolve stalled replication forks, the accumulation of DNA damage and rapid cell death (32, 33).While normal cells can generally tolerate inhibition of ATR by activating compensatory DNA repair pathways, such pathways are frequently defective in cancer cells, rendering them highly dependent on ATR for survival. Due to its major implication in RS-induced DDR pathway activation, ATR has been recently considered as a potential target in various cancer models and several ATR inhibitors are under clinical evaluation. Classically, tumors with high level of RS have been suggested to be the most sensitive to ATR inhibitors, including RS-induced by oncogenic amplification such as MYC, RAS or Cyclin E1. Other potential molecular alterations that may sensitize to ATR inhibitors are those associated with HRD (33, 34) as well as those associated with DDR such as loss of expression of ATM, ARID1A, ERCC4, XRCC1, RB133, (35-39). Of note, recent works have revealed that treatment with ATR inhibitors can overcome the resistance to PARP inhibition (40), suggesting the potential of ATR inhibitors as a second-line treatment in patients who have developed resistance to PARP inhibitors (33).

ATR inhibitors and M1774:

First early-phase studies have been initiated using ATR inhibitors as monotherapy or in combination with various therapeutics including chemotherapy and PARP inhibitors in various tumor types. Tolerance was favorable and preliminary proofs of activity have been obtained, notably in patients with DDR and/or HR pathway alterations (41-43). M1774 (substance code MSC2584415A; also known as VXc-400 or VRT-1363004) is an orally administered small molecule inhibitor of ATR kinase; it is a potent and selective inhibitor of ATR, with a mean half maximal inhibitory concentration (IC50) of 4 nM, as measured by inhibition of the phosphorylation of the proximal target CHK1 in cells (M1774's IB V2.0, Nov 2020). Pre-clinical pharmacology, pharmacokinetic (PK), and toxicology studies support development of M1774 for the treatment of patients with advanced cancers and a phase I study is currently ongoing.

As of 21 APR 2022, 55 participants received doses of M1774 ranging from 5 mg to 270 mg once daily (QD). Dose-limiting toxicities (DLT) were observed at dose levels of 130 mg QD and above. DLT included grade 2 and 3 anemia requiring transfusion in 7 patients, as well as one grade 4 thrombopenia associated with upper gastro-intestinal hemorrhage. Most frequent toxicities also included gastro-intestinal disorders (nausea, vomiting, constipation, diarrhea and abdominal pain). The recommended phase 2 dose as monotherapy was 180 mg QD, 2 weeks on/ 1 week off. Of note, preliminary data showed that PK was approximately dose proportional up to 180 mg and slightly more than dose proportional beyond 180 mg. Absorption was fast with median Tmax ranging from 1 to 3.5 hours and mean T1/2 ranged from 3 to 5.6 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age (or > 18, depending on countries' legal age of majority) at the time of signing the informed consent.
2. Man or postmenopausal woman due to either surgical/natural menopause or chemical ovarian suppression (maintained during all the study treatment) with a gonadotropin-releasing hormone (GnRH) agonist or radiation-induced ovarian suppression.
3. Patient has advanced (loco regionally recurrent not amenable to curative therapy or metastatic) breast cancer.
4. Patient has pathologically confirmed hormone receptors (HR)-positive (ER+ and/or PgR+) and HER2-negative advanced BC by local laboratory on the last tissue examined. HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing
5. Patient has disease progression while receiving aromatase inhibitor therapy (i.e. letrozole, anastrozole, exemestane) in combination with CDK4/6 inhibitors (palbociclib, ribociclib, abemaciclib) administered in the advanced setting or patients has recurrence while receiving aromatase inhibitor therapy (i.e. letrozole, anastrozole, exemestane) in combination with CDK4/6 inhibitors (palbociclib, ribociclib, abemaciclib) or within 12 months of the end of CDK4/6 inhibitors when administered in the early setting.
6. For phase 2 part only : patient whose tumor displays (according to local tumor boards) either

   * Germline or somatic BRCA1, BRCA2 or PALB2 mutations and prior exposure and resistance to PARP inhibitors (cohort 1).
   * Documented deleterious germline or somatic alterations associated with HRD : BARD1 BRIP1, CDK12, CHEK2, FANCA, FANCD2, FANCL, MRE11A, NBN, PPP2R2A, RAD51B, RAD51C, RAD51D and RAD54L (cohort 2). Patients with sBRCA1, sBRCA2 and g/sPALB2, without previous exposure to PARP inhibitors, may be enrolled in this cohort.
   * Oncogenic driver amplification (such as MYC, RAS, Cycin E1) or mutations of the following genes: ATM, ARID1A, ERCC4, XRCC1, RB1, ATRX, DAXX, suspected to favor RS and thereby sensitivity to ATR inhibitors as determined by a local molecular tumor board and validated by the central molecular tumor board (cohort 3).
7. Tumor site accessible for baseline biopsy or archival tissue available without any specific anticancer treatment after collection
8. No more than one previous chemotherapy regimen for advanced disease (including antibody drug conjugates) ; (neo)adjuvant chemotherapy is allowed
9. No more than 1 previous endocrine therapy administered for metastatic disease
10. Patient with gBRCA1/2 must have received PARP inhibitors and have experienced disease progression during or after treatment
11. Patient has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
12. Patient must have normal organ and marrow function

    Adequate hematologic function as indicated by:
    * Platelet count ≥ 100,000/mm3
    * Absolute neutrophil count > 1,500/µL with no growth factor treatment within the last 14 days
    * Hemoglobin ≥ 10.0 g/dL, with no erythropoietin or red blood cell transfusion within the last 14 days.

    Adequate hepatic function as indicated by:
    * Total bilirubin ≤ 1.5 × ULN. In the case of documented Gilbert's syndrome, total bilirubin ≤ 2.0 × ULN is allowed.
    * AST and ALT levels ≤ 3 × ULN or ≤ 5 × ULN in presence of liver metastases.
13. Adequate renal function defined as: serum creatinine ≤ 1.5 × ULN. If serum creatinine is > 1.5 × ULN, creatinine clearance needs to be ≥ 60 mL/min by calculation using the Cockcroft-Gault formula or by measured 24-hour urine collection. The Cockcroft-Gault formula is (glomerular filtration rate [mL/min] = {(l40-age) × weight/(72 × serum creatinine [mg/dL])} × 0.85 [if female]).
14. A female participant must have a negative serum pregnancy test, as required by local regulations, before the first dose of study intervention).

    Contraceptive use will be consistent with local regulations on contraception methods for those participating in clinical studies.

    Female participants of childbearing potential will be using highly effective contraception for throughout the study and for at least 6 months after last M1774 treatment administration. Women should not breastfeed during the study and for at least 1 month after the study period, (i.e., after the last dose of study intervention is administered).

    Male participants will be using highly effective contraception for throughout the study and for at least 3 months after last M1774 treatment administration.
15. Patient has measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria
16. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen or any other regimen of social security
17. Are capable of giving signed informed consent(or a trusted person) , which includes compliance with the requirements and restrictions listed in the ICF and this protocol.

Exclusion Criteria:

1. Has received previous fulvestrant
2. Any investigational therapy within ≤ 21 days or 5 half-lives prior treatment, whichever is longer, prior treatment
3. Any hormonal therapy within 7 days prior treatment (except ovarian function suppression).
4. Any cytotoxic therapy within 21 days (3-weekly regimen), 14 days (weekly or oral regimen) prior treatment
5. Previous treatment with ATR or CHK1 inhibitors (unless treatment was for less than 3 weeks duration and at least 12 months have elapsed between the last dose and randomization. Patients that did not tolerate prior treatment are excluded). Prior treatment with PARP inhibitor is allowed
6. . .
7. Patients with second primary cancer, EXCEPTIONS: adequately treated non melanoma skin cancer, curatively treated in-situ cancer of the cervix, Ductal carcinoma in Situ (DCIS), stage 1 grade 1 endometrial carcinoma, or other solid tumours curatively treated with no evidence of disease for ≥ 3 years prior to study entry (including lymphomas [without bone marrow involvement]).
8. Mean resting corrected QTc interval using the Fridericia formula (QTcF) = >470 msec/female patients and >450 msec for male patients obtained from 3 ECGs Uncontrolled or poorly controlled arterial hypertension, symptomatic congestive heart failure (New York Heart Association Classification ≥ Class III), uncontrolled cardiac arrhythmia, calculated QTc average using the QTcF > 470 msec; unstable angina pectoris, myocardial infarction or a coronary revascularization procedure, cerebral vascular accident, transient ischemic attack, or any other significant vascular disease within 180 days of study intervention start.
9. Any of the following cardiac diseases currently or within the last 6 months
10. Unstable angina pectoris
11. Congestive heart failure ≥ Class 2 as defined by the New York Heart Association
12. Acute myocardial infarction
13. Conduction abnormality not controlled with pacemaker or medication (patients with a conduction abnormality controlled with pacemaker or medication at the time of screening are eligible)
14. Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
15. Other clinically significant heart disease
16. Concomitant use of known strong cytochrome P (CYP) 3A inhibitors (eg itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem,fluconazole, verapamil).
17. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil).
18. Persistent toxicities (≥ CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and CTCAE grade 2 peripheral neuropathy.
19. Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
20. Immunocompromised patients, eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
21. Patients with known active hepatitis (ie, hepatitis B or C).
22. Visceral crisis or impending visceral crisis at time of screening.
23. CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement).
24. uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, or severe malnutrition.
25. Active infection requiring antibiotics at day 1 of cycle 1
26. Active and/or uncontrolled infection. The following exceptions apply:

    * Participants with HIV infection are eligible if they are on effective antiretroviral therapy with undetectable viral load within 6 months, provided there is no expected drug-drug interaction.
    * Participants with evidence of chronic HBV infection are eligible if the HBV viral load is undetectable on suppressive therapy (if indicated), and if they have ALT, AST, and total bilirubin levels < ULN, and provided there is no expected drug-drug interaction.
    * Participants with a history of HCV infection are eligible if they have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load, and if they have ALT, AST, and total bilirubin levels < ULN.
27. Participants with clinically controlled brain metastases, which is defined as individuals with central nervous system metastases that have been treated for, are asymptomatic, and have discontinued corticosteroids for > 14 days or are on a stable or decreasing steroid dose (for the treatment of brain metastases) may be enrolled. Participants with meningeal carcinomatosis are excluded.
28. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease (SD) for 28 days.
29. Patients with a history of treated central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria: Disease outside the CNS is present. No clinical evidence of progression since completion of CNS-directed therapy. Minimum of 3 weeks between completion of radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥3) acute toxicity with no ongoing requirement for >10 mg of prednisone per day or an equivalent dose of other corticosteroid. If on corticosteroids, the patient should be receiving a stable dose of corticosteroids, started at least 4 weeks prior to treatment
30. Any other clinical condition, uncontrolled concurrent illness, or other situations, which in the Investigator's opinion would not make the patient a good candidate for the study or may potentially impact the absorption of M1774 such as (but not limited to) significant small bowel resection, gastric surgery, or exocrine pancreatic insufficiency requiring pancreatic enzyme replacement therapy.
31. Live vaccines within 4 weeks of first dose of study intervention and while receiving study intervention. Administration of inactivated vaccines (i.e., inactivated influenza vaccine) is permitted. Inactivated RNA or nonreplicating viral vector-based SARS-CoV-2 vaccines are allowed, as approved by local/regional Health Authorities. Novel live attenuated SARS CoV-2 vaccines are not permitted.
32. Persistence of AEs related to any prior treatments that have not recovered to Grade ≤ 1 unless AEs are clinically non significant (e.g. alopecia) and /or stable on supportive therapy in the opinion of the Investigator.
33. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
34. History or known hypersensitivity to the active substances or to any excipients of the study interventions.
35. Pregnant or breast feeding women.
36. Patient considered socially or psychologically unable to comply with the treatment and the required medical follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity | 28 days after the first dose of treatment
  incidence of dose-limiting toxicity as defined as considered to be related or possi-bly related to M1774 or fulvestrant treatment

SECONDARY OUTCOMES:
Tolerance | 18 months after the first dose of treatment
  incidence of AEs and Serious Adverse Events (SAE) presented by grade according to the NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No